CLINICAL TRIAL: NCT03050905
Title: An Open-Label, Proof of Concept Study To Evaluate the Efficacy and Justification Of OBV/PTV/r and DSV In Adults With Chronic Hepatitis C Virus (HCV) Infection Genotype 2K/1B- NINJA Study
Brief Title: Proof of Concept Study To Evaluate the Efficacy and Justification Of OBV/PTV/r and DSV In Adults With Chronic Hepatitis C Virus Genotype 2K/1B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NINJA Study - 11227
Record Dates: First submitted 2016-12-11; First posted 2017-02-13 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: HCV Coinfection
MeSH Terms: interventions — dasabuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The study will include 1 group. Patients will be treated according to label recommendation as for GT1b (with and without cirrhosis) for 12 weeks. All subjects will receive Ombitasvir+Paritaprevir+Ritonavir (VEKIRAX) and Dasabuvir (EXVIERA).
  Interventions: Drug: VEKIRAX; Drug: EXVIERA

INTERVENTIONS:
Drug: VEKIRAX — Patients will be treated according to label recommendation as for GT1b (with and without cirrhosis) for 12 weeks. All subjects will receive Ombitasvir+Paritaprevir+Ritonavir (Viekirax).
  Study Regimen: ombitasvir+paritaprevir+ritonavir (25+150+100mg once daily)
  Other Names: Ombitasvir+Paritaprevir+Ritonavir
Drug: EXVIERA — Patients will be treated according to label recommendation as for GT1b (with and without cirrhosis) for 12 weeks. All subjects will receive Dasabuvir (Exviera).
  Study Regimen: dasabuvir (250 mg twice daily)
  Other Names: Dasabuvir

SUMMARY:
HCV infection is one of the most prevalent etiologies for liver cirrhosis and hepatocellular carcinoma. HCV is highly heterogeneous, with seven confirmed major genotypes. Each genotype displays a different geographic distribution.

Since different HCV genotypes react differently on available antiviral therapies, the correct identification of HCV genotype serves as a marker of responsiveness and an indicator for duration of treatment.

The recombinant HCV genotype 2k/1b was first described in Saint Petersburg in 2002.

A sequencing strategy led to the detection of HCV genotype 2k/1b. However, clinical laboratories often use the VERSANT HCV Genotype 2.0 Assay for routine HCV genotyping. This assay may potentially misclassify these HCV strains as genotype 2a/2c. Based on these findings, the number of patients with 2k/1b may be underestimated.

AbbVie's IFN-free regimen for the treatment of chronic HCV genotype 1b infection includes 3 DAAs with distinct mechanisms of action and non-overlapping resistance pattern to target HCV proteins essential for viral replication. The high efficacy of the 3D regimen was proven in registration clinical trials and RW for 1b population.

3D regimen has not been evaluated for patients with HCV genotype 2K/1B. Primary Objective

• Evaluate the efficacy of ombitasvir/paritaprevir/ritonavir and dasabuvir (3D) in an interferon-free treatment regimen as assessed by SVR in adult patients with HCV 2k/1b.

Study Design:

.The study will include 1 group. Patients with HCV GT 2k1b will be treated according to label recommendation as for GT1b (with and without cirrhosis) for 12 weeks. All subjects will receive Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir. Subjects will be assessed for antiviral response, clinical outcomes, patient reported adverse events and presence and emergence of resistance associated variants. Subjects will be followed for up to 12 weeks of treatment and extra 24 weeks of follow up. Scheduled visits will include: physician assessment and blood tests including HCV resistance mutations.

DETAILED DESCRIPTION:
Study Procedures:

Initial screening period:

HCV GT2K/1B -infected subjects who will be meeting eligibility criteria, will provide written informed consent, perform baseline RAS testing and will be enrolled to the study.

Baseline period:

On day 0, all patients will be assessed by a general physical examination, blood and urine tests including HCV resistance mutations (elaborated in the budget file), Fibroscan or SHEAR WAVE Elastography and abdominal ultrasound. After the initial assessment all included will be allocated for treatment.

Study configuration:

The study will include 1 group of patients infected GT 2k1b. Patients will be treated according to label recommendation for GT1b (with and without cirrhosis) for 12 weeks. All subjects will receive Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir. Scheduled visits will take place in 0, 4, 12 and 24 weeks for all patients.

All visits will include: physician assessment and blood tests as elaborated in the Study Flowchart. Subjects will be assessed for antiviral response, clinical outcomes, patient reported adverse events and presence and emergence of resistance associated variants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male and female
* HCV Genotype 2K/1B (P/R experienced or naïve; non-cirrhotic/ Comp. cirrhotic CP-A 5)
* Capable to provide informed consent

Exclusion Criteria:

* Could not remain in the study for 36 weeks
* Co-infected with human immunodeficiency virus (HIV) or HBV
* Severe renal impairment (calculated creatinine clearance <30 mL/min )
* Evidence of hepatocellular carcinoma (HCC)
* Severe concurrent disease
* Pregnant, lactating, expecting to conceive or donate eggs or male participant with pregnant female partner
* DAA treatment experienced
* History of drug or alcohol abuse within 6 months prior enrolment - positive result of a urine drug screen at the screening visit and a positive result on the alcohol consumption questioner.
* Evidence or history of chronic liver disease not caused by HCV Participants currently enrolled in an HCV-related research protocol OR currently receiving HCV treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
The percentage of patients achieving SVR12 (single last HCV RNA <12 IU/mL 12 weeks after the last actual dose of the ABBVIE regimen) | 12 weeks post treatment

SECONDARY OUTCOMES:
Safety: absolute and relative numbers of discontinuations, AE and SAEs (Number of Participants With Adverse Events That Are Related to Treatment). | 36 weeks
Resistance Associated Substitute (RAS): The percentage of patients with the presence of RAS's- at baseline and at post-treatment weak 12. | 12 weeks post treatment
Time of virologic failure using population sequencing; SVR12 rate | 36 weeks
Time of virologic failure using population sequencing; presence of BL RAS's. | 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided